CLINICAL TRIAL: NCT07226947
Title: BIA Monitoring and Exercise for the Prevention of Muscle Loss With Incretin Therapy (BICEP Study)
Brief Title: Body Composition and Exercise to Prevent Muscle Loss With GLP1 Agonist Treatment
Acronym: BICEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Samsung (Industry)
Responsible Party: Principal Investigator, Melissa Susan Putman, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025P001490
Record Dates: First submitted 2025-11-06; First posted 2025-11-12 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Body Composition
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartwatch activity monitor (Experimental): Participants will be provided a smartwatch to monitor activity and body composition monitor. They will also have exercise goals set with reminders on the watch.
  Interventions: Device: Smartwatch activity and body composition monitor; Behavioral: General guidance on recommended exercise
- Usual guidance (Active Comparator): Participants will receive general guidance on recommended exercise
  Interventions: Behavioral: General guidance on recommended exercise

INTERVENTIONS:
Device: Smartwatch activity and body composition monitor — Participants will be provided a smartwatch to monitor their exercise and body composition
  Arms: Smartwatch activity monitor
Behavioral: General guidance on recommended exercise — Participants will receive general guidance on recommended exercise

SUMMARY:
The goal of this study is to learn if a smartwatch that measures activity level and body composition, combined with exercise reminders, can safely improve strength and muscle mass in people who recently started or are planning to start treatment with incretin therapy (liraglutide, semaglutide, tirzepatide or retatrutide), also known as glucagon-like peptide 1 receptor agonist (GLP-1 RA) medications.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years old at time of signing informed consent
2. Started treatment with incretin therapy (liraglutide, semaglutide, tirzepatide, or retatrutide) within the past 2 months or planning to start this treatment

   a. Potential participants switching GLP1-RA therapies due to inadequate response to a prior treatment will be eligible for enrollment
3. Able to provide informed consent

Exclusion Criteria

1. Current pregnancy (positive urine hCG) or plans to become pregnant in the next 6 months
2. BMI <25 kg/m2 at the time of screening
3. Unable to participate in a regular physical exercise program
4. Implanted pacemaker
5. Any factors that, in the opinion of the principal investigator, would interfere with the safe completion of the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Lean mass (kg) | 6 months
  Dual-energy X-ray absorptiometry (DXA) body composition measure

SECONDARY OUTCOMES:
Lean mass index (kg/m2) | 6 months
  Dual-energy X-ray absorptiometry (DXA) body composition measure
Appendicular lean mass index (kg/m2) | 6 months
  Dual-energy X-ray absorptiometry (DXA) body composition measure
Fat mass index (kg/m2) | 6 months
  Dual-energy X-ray absorptiometry (DXA) body composition measure
Fat mass (kg) | 6 months
  Dual-energy X-ray absorptiometry (DXA) body composition measure
Visceral adipose tissue (kg) | 6 months
  Dual-energy X-ray absorptiometry (DXA) body composition measure
Lean mass/fat mass ratio | 6 months
  Dual-energy X-ray absorptiometry (DXA) body composition measure
Fat free mass | 6 months
  Bioimpedance analysis body composition measure
Hand grip strength (kg) | 6 months
  Function strength measurement
1-minute sit-to-stand | 6 months
  Number of sit-to-stand repetitions in one minute
6-minute walk test | 6 months
  Distance walked in six minutes
Short Physical Performance Battery frailty score (total points) | 6 months
  Physical functioning test consisting of standing balance, gait speed, and repeated chair stands
Physical activity score | 6 months
  International Physical Activity Questionnaire (IPAQ)

OTHER OUTCOMES:
Lumbar spine bone mineral density (g/cm2) | 6 months
  Dual energy Xray absorptiometry
Total hip bone mineral density (g/cm2) | 6 months
  Dual energy Xray absorptiometry
Femoral neck bone mineral density (g/cm2) | 6 months
  Dual energy Xray absorptiometry
Dimensional Anhedonia Scale (DARS) | 6 months
  17 item Self-report scale that measures anhedonia, scores measured from 0-68 with higher scores signifying a better outcome.
Patient Health Questionaire-8 (PHQ-8) | 6 months
  8-item scale that measures depressive symptoms over the past two weeks
Generalized Anxiety Disorder 7 item scale (GAD-7) | 6 months
  7-item scale that measures anxiety symptoms over the past few days. Scores measured from 0-21 with higher scores signifying a worse outcome.
Participant feedback survey | 6 months
  Survey with questions to understand participant experience with the study

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Putman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Diabetes Research Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.

REFERENCES:
- [Background] Locatelli JC, Costa JG, Haynes A, Naylor LH, Fegan PG, Yeap BB, Green DJ. Incretin-Based Weight Loss Pharmacotherapy: Can Resistance Exercise Optimize Changes in Body Composition? Diabetes Care. 2024 Oct 1;47(10):1718-1730. doi: 10.2337/dci23-0100. PMID 38687506
- [Background] Cesari M, Leeuwenburgh C, Lauretani F, Onder G, Bandinelli S, Maraldi C, Guralnik JM, Pahor M, Ferrucci L. Frailty syndrome and skeletal muscle: results from the Invecchiare in Chianti study. Am J Clin Nutr. 2006 May;83(5):1142-8. doi: 10.1093/ajcn/83.5.1142. PMID 16685058
- [Background] Srikanthan P, Horwich TB, Tseng CH. Relation of Muscle Mass and Fat Mass to Cardiovascular Disease Mortality. Am J Cardiol. 2016 Apr 15;117(8):1355-60. doi: 10.1016/j.amjcard.2016.01.033. Epub 2016 Feb 2. PMID 26949037
- [Background] Tyrovolas S, Haro JM, Mariolis A, Piscopo S, Valacchi G, Bountziouka V, Anastasiou F, Zeimbekis A, Tyrovola D, Foscolou A, Gotsis E, Metallinos G, Tur JA, Matalas A, Lionis C, Polychronopoulos E, Panagiotakos D. Skeletal muscle mass and body fat in relation to successful ageing of older adults: The multi-national MEDIS study. Arch Gerontol Geriatr. 2016 Sep-Oct;66:95-101. doi: 10.1016/j.archger.2016.04.017. Epub 2016 May 9. PMID 27266673
- [Background] Tempia Valenta S, Nicastri A, Marcolini F, Petroni ML, Perazza F, Beghelli V, et al. The Impact of GLP-1 Receptor Agonists (GLP-1 RAs) on Mental Health: A Systematic Review. Current Treatment Options in Psychiatry. 2024 Sep 18;11(4):310-57.
- [Background] Jastreboff AM, Kaplan LM, Frias JP, Wu Q, Du Y, Gurbuz S, Coskun T, Haupt A, Milicevic Z, Hartman ML; Retatrutide Phase 2 Obesity Trial Investigators. Triple-Hormone-Receptor Agonist Retatrutide for Obesity - A Phase 2 Trial. N Engl J Med. 2023 Aug 10;389(6):514-526. doi: 10.1056/NEJMoa2301972. Epub 2023 Jun 26. PMID 37366315
- [Background] Garvey WT, Frias JP, Jastreboff AM, le Roux CW, Sattar N, Aizenberg D, Mao H, Zhang S, Ahmad NN, Bunck MC, Benabbad I, Zhang XM; SURMOUNT-2 investigators. Tirzepatide once weekly for the treatment of obesity in people with type 2 diabetes (SURMOUNT-2): a double-blind, randomised, multicentre, placebo-controlled, phase 3 trial. Lancet. 2023 Aug 19;402(10402):613-626. doi: 10.1016/S0140-6736(23)01200-X. Epub 2023 Jun 26. PMID 37385275
- [Background] Jastreboff AM, Aronne LJ, Ahmad NN, Wharton S, Connery L, Alves B, Kiyosue A, Zhang S, Liu B, Bunck MC, Stefanski A; SURMOUNT-1 Investigators. Tirzepatide Once Weekly for the Treatment of Obesity. N Engl J Med. 2022 Jul 21;387(3):205-216. doi: 10.1056/NEJMoa2206038. Epub 2022 Jun 4. PMID 35658024
- [Background] Wilding JPH, Batterham RL, Calanna S, Davies M, Van Gaal LF, Lingvay I, McGowan BM, Rosenstock J, Tran MTD, Wadden TA, Wharton S, Yokote K, Zeuthen N, Kushner RF; STEP 1 Study Group. Once-Weekly Semaglutide in Adults with Overweight or Obesity. N Engl J Med. 2021 Mar 18;384(11):989-1002. doi: 10.1056/NEJMoa2032183. Epub 2021 Feb 10. PMID 33567185
- See also: Recruitment website for this study — https://rally.massgeneralbrigham.org/study/bicepstudy